CLINICAL TRIAL: NCT05035758
Title: Transcendental Meditation and Yoga: Short- and Long-term Effects in Cardiac Rehabilitation Patients - a Pilot Study
Acronym: TMY_Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EK 31-443 ex 18/19
Record Dates: First submitted 2021-08-19; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Vascular Diseases; Stress, Psychological
MeSH Terms: conditions — Cardiovascular Diseases; Vascular Diseases; Stress, Psychological | interventions — Meditation; Yoga

STUDY DESIGN:
Intervention Model Description: In this study, we will separate the patients into three groups; the control group (A) receives the standard exercise therapy that is part of the rehabilitation at the center. The intervention group B additionally to this standard therapy receives transcendental meditation sessions. Intervention group C also receives the standard rehabilitation exercise training and in addition yoga sessions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Goups (No Intervention): The control group (A) receives standard exercise therapy that is part of the rehabilitation at the center and no additional intervention
- Transcendental Meditation (Experimental): The intervention group (B) receives transcendental meditation sessions (twice per day for 30 minutes) additionally to the standard rehabilitation therapy.
  Interventions: Other: Transcendental Meditation
- Yoga (Experimental): The intervention group (C) receives yoga sessions (twice per day for 30 minutes) additionally to the standard rehabilitation therapy.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Transcendental Meditation — In the beginning, the patients from group B will receive an introductory lecture about transcendental meditation (TM) which includes general information, the procedure itself and other techniques of relaxation and personal development.
  In this first session the method is learned by practice, in the following 3 meetings additional instructions are given about the correct practice of the TM technique; TM is practiced twice a day for 20 minutes. The method is easy to learn and effortless. To guarantee the right performance of TM by the patients, there will be two group meetings per week and one individual personal meeting with the TM teacher.After discharge from the rehabilitation program (after 4 weeks) there will be meetings offered according to the patients need. This will then be arranged individually.
  Arms: Transcendental Meditation
Other: Yoga — In addition to the standard rehabilitation exercise training, the patients in this group will receive a 20-minute workshop where they learn how to do the yoga exercise. The initial yoga workshop will be held by Dr. Gilda Wüst who is a yoga expert with a lot of experience based in St. Radegund.
  After this, yoga sessions will be included (additionally to the regular/standard exercise) into their daily timetable. Two yoga sessions will be done every day, one in the morning (6:30-6:50) and one in the evening (16:30-16:50) and will last for about 20 minutes.
  Arms: Yoga

SUMMARY:
Atherosclerotic cardiovascular disease (CVD) is the leading cause of death in Austria. The ESC guidelines recommend cardiac rehabilitation after coronary events (acute coronary syndrome, myocardial infarction, etc) with the highest level of evidence. Drug therapy and non-pharmacological measures such as a targeted and individualized exercise program, stress management programs, reduction of cardiovascular risk parameters through training, nutritional counseling, smoking cessation, etc. reduce the cardiovascular risk of recurrence. The reduction of psychosocial stress is regarded as one of the major factors in cardiac rehabilitation, alongside physical training and nutrition.

In this study, transcendental meditation (TM) and yoga will be added on top of regular cardiac rehabilitation to investigate the efficiency of these methods to possibly improve the quality of life of recovering patients. Both methods are believed to reduce stress for users, while being relatively easy to introduce to and implement in daily life for beginners, carrying no extra cost for them further down the line. The main hypothesis is that cardiac patients undergoing rehabilitation plus TM or yoga therapy will show changes in endothelial function, micobiome and stress levels. Three groups of 10 participants from a cardiac cardiac rehabilitation will be subjected to standard rehabilitation, rehabilitation with meditation, and rehabilitation with yoga, respectively. The vascular state of each patient will be closely monitored over the 4 weeks, as well as after a 1-year follow up. Furthermore, the expected stress reductions will be assessed in short term and long-term by researching hair cortisol levels, on top of self-reporting questionnaires.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (CVD) is the leading cause of death in Austria. The ESC guidelines recommend cardiac rehabilitation after coronary events (acute coronary syndrome, myocardial infarction, etc) with the highest level of evidence. Drug therapy and non-pharmacological measures such as a targeted and individualized exercise program, stress management programs, reduction of cardiovascular risk parameters through training, nutritional counseling, smoking cessation, etc. reduce the cardiovascular risk of recurrence. Patients following coronary events will be eligible for in-patient rehabilitation after the acute events at the Rehabilitation Center of the Pensionsversicherungsanstalt in St. Radegund near Graz. The rehabilitation center with 150 beds is located at an altitude of 717m in the spa town of St. Radegund near the provincial capital of Graz at the foot of the Schöckl.

Substantial epidemiological and mechanistic research has demonstrated that psychosocial stress contributes to CVD pathophysiology and clinical events. However, there is paucity of clinical trial data on the effects of stress reduction on cardiovascular clinical events. The reduction of psychosocial stress is regarded as one of the major goals in cardiac rehabilitation, in addition to encouraging exercise and improved nutrition (Yusuf et al., 2004). Meditation and Yoga are two different methods that can be performed to increase mindfulness and reduce stress.

1. Transcendental Meditation (TM) Previous controlled clinical studies have reported that a selected stress reduction technique, the Transcendental Meditation program (TM) is associated with reductions in CVD risk factors. These include hypertension, insulin resistance, cigarette smoking, reduced CVD events such as stroke and heart attack, and reduced psychosocial stress and surrogate markers of disease such as carotid intima-media thickness, left ventricular mass and stress-induced myocardial ischemia. TM is also believed to lead to a higher EEG coherence.

   The procedure of Transcendental Meditation (TM) is a technique with a millennia-old tradition. For more than 50 years, specially trained and authorized transcendental meditation teachers as directed by vedic teacher Maharishi Mahesh Yogi have taught it worldwide. It is not coupled to a system of religion (Hinduism, Buddhism, etc.), nor is it bound to particular beliefs, intellectual abilities, concentration, physical or mental condition.

   The TM technique is described as a simple, natural, effortless procedure that is practiced 20 minutes twice a day while sitting comfortably with eyes closed. During the practice, it is reported that ordinary thinking processes settle down, and a distinctive wakeful hypometabolic state characterized by neural coherence and physiological rest is achieved. During the practice of TM, the mind effortlessly and systematically experiences finer stages of thought and eventually transcends the finest mental impulse to experience a state of restful wakefulness, the ground state of consciousness.

   The technique of TM is a distinct, well-defined meditation program that differs fundamentally from all other methods of concentration and contemplation. According to scientific studies, three basic mechanisms of meditation are distinguished:
   * Concentrative Attention Techniques
   * mindfulness techniques
   * automatically self-transcending techniques

   The technique of Transcendental Meditation is the main representative of this last group. It is practiced twice daily for 15-20 minutes. You sit comfortably on a chair and have your eyes closed. During the process of TM meditation, the mind becomes silent, but remains fully awake. It allows to achieve a deep relaxation of mind and body. Due to its simplicity and efficiency, the technique of transcendental meditation is particularly suitable for use in the field of preventive medicine and health education.
2. Yoga Yoga originated in India thousands of year ago. The practice of yoga unifies the mind and body through coordinated breathing (pranayama), movement (asana), and meditation (dhyana), which has been known to promote well-being and reduce stress. In the last several decades, the millions of practitioners and the rise of yoga studios have popularized yoga in the western society.

Yoga is a form of mind-body fitness that involves a combination of muscular activity and an internally directed mindful focus on awareness of the self, breath, and energy. It aims at developing an integrated personality, where the growth of physical, mental, social, and spiritual planes is equally focused. The advantage of yoga is that its benefits are available to a wide range of people, from young to elderly, healthy or sick.

Yoga has shown promising results in different publications as both an intervention and a rehabilitation mean, particularly as an element of lifestyle change for cardiac patients. Trials have been run for patients post MI and stroke, and while conclusive evidence is necessary to confirm the feasibility of the proposed methods, yoga has been also used by patients with heart failure (all classes), and hypertension.

Although several studies evaluated effects of Transcendental Meditation (TM) and Yoga, effects like endothelial function changes, as well as the influence of TM and/or Yoga on the physiological functions including vascular function, intima-media thickness of the arteries, the gut microbiome and gut barrier function in context of inflammatory parameters have been relatively less investigated. Less is known about the effects of TM and Yoga on outcome parameters in rehabilitation patients, undergoing 4 weeks of cardiac rehabilitation as well. The purpose of this study is to investigate whether interventions such as TM or Yoga during inpatient cardiac rehabilitation, in addition to the standard rehabilitation therapy, can provide additional benefits in terms of lowering the cardiac risk parameters.

Aim of the study The overarching aim of this project is to explore how TM or yoga, applied in addition to the existing exercise protocol , affects the physiological functions of blood vessels (arterial and venous) as well as autonomic function and stress levels. Supine to stand test will be carried out to assess how autonomic function is altered with treatment. Flow mediated dilatation, intima media thickness, pulse wave velocity and retinal imaging will be done to assess the vascular state of each patient over the four weeks of rehabilitation and after a one-year follow up. Finally, the stress reductions with TM will be assessed in short term and long-term using measurements of hair cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients after myocardial infarction (MI)
* after ST-level myocardial infarction (STEMI) and
* non ST-level myocardial infarction (NSTEMI)
* after acute coronary syndrome (ACS)
* coronary artery disease (CAD) with percutaneous coronary intervention (PCI),
* after coronary artery bypass graft (CABG)
* age range 40-80
* admitted to the cardiac rehabilitatoin center in St. Radegund.

Exclusion Criteria:

* patients who must be monitored because of clinical symptoms (subjects with NYHA III, mini mental score more than 26, or subjects who are not sufficiently mobilized)
* subjects who regularly perform Yoga exercises or any other meditation techniques

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of arterial Stiffness | through study completion, an average of 1 year
  Arterial Stiffness will be assessed using pulse wave velocity measurement via the vicorder device
Change of Retinal Microvasculature | through study completion, an average of 1 year
  Will be assessed via retinal imaging
Changes in heart rate to orthostatic loading | through study completion, an average of 1 year
  Patients will be asked to sit for 5 minutes and then stand up straight for 5 minutes. Changes in heart rate during this period will be assessed.
Changes in blood pressure to orthostatic loading | through study completion, an average of 1 year
  Patients will be asked to sit for 5 minutes and then stand up straight for 5 minutes. Changes in blood pressure during this period will be assessed.
Changes in Microbiome Samples | through study completion, an average of 1 year
  Stool samples will be collected to analyse the changes in the microbiome
Change in stress levels via cortisol measurements from hair samples | through study completion, an average of 1 year
  Hair samples will be collected from the posterior vertex and cut as close to the scalp as possible and cut in pieces with 1 cm each. 1 cm equals 1 month of stress levels. A minimum of 10 mg of hair will be used for each sample.
Changes in The Pittsburgh Sleep Quality Index (PSQI) | through study completion, an average of 1 year
  self-report questionnaire that assesses sleep quality over a 1-month time interval
Changes in SF-36 | through study completion, an average of 1 year
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.
Changes in POMS - short form | through study completion, an average of 1 year
  POMS measures six different dimensions of mood swings over a period of time. These include: Tension or Anxiety, Anger or Hostility, Vigor or Activity, Fatigue or Inertia, Depression or Dejection, Confusion or Bewilderment.
Changes in PSQ20 | through study completion, an average of 1 year
  The aim of the Perceived Stress Questionnaire is to identify and investigate the subjective perception, evaluation and further processing of stressors. This should also question the dominance and objectivity of external stressors.
Changes in Spielberger State Trait Anxiety Inventory (STAI) | through study completion, an average of 1 year
  It consists of two parts (each 20 questions) rating the answers on a 4-point scale. The score for the global test may range between 40-160 points. It evaluates state anxiety (in a specific situation) or trait anxiety (as part of a person´s character).
Changes in Tryptophan pathway | through study completion, an average of 1 year
  Tryptophan as stress marker from plasma samples
Changes in Kynurenin levels | through study completion, an average of 1 year
  Kynurenin as stress marker from plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Nandu Goswami, MD, Principal Investigator — nandu.goswami@medunigraz.at
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided